CLINICAL TRIAL: NCT03493360
Title: Feedback Visual na Lombalgia crónica da grávida e da não grávida/ Visual Feedback in Chronic Low Back Pain of Pregnant and Nonpregnant Women
Brief Title: Visual Feedback in Chronic Low Back Pain of Pregnant and Nonpregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-CED/2018
Record Dates: First submitted 2018-04-04; First posted 2018-04-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Feedback, Sensory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual feedback (Experimental): Participants will be asked to perform movements of the low back while looking at a mirror for visual feedback.
  Interventions: Other: Visual feedback
- No visual feedback (Active Comparator): Participants will be asked to perform movements of the low back while the mirrors are covered and no visual feedback is provided.
  Interventions: Other: No visual feedback

INTERVENTIONS:
Other: Visual feedback — Participants will be asked to perform 10 repetitions of low back flexion, extension and lateral side-flexions while looking at their back in a mirror for visual feedback.
  Arms: Visual feedback
Other: No visual feedback — Participants will be asked to perform 10 repetitions of low back flexion, extension and lateral side-flexions while looking at a mirror that is covered and no visual feedback is provided.
  Arms: No visual feedback

SUMMARY:
The objectives of this study are to:

* Evaluate the effect of visual feedback on the intensity of low back pain, range of motion and function of pregnant and non-pregnant women with chronic low back pain.
* Determine the association between low back pain, catastrophizing, fear of movement and low back perception/image.

DETAILED DESCRIPTION:
It is antecipated that 15 pregnant women with low back pain and 15 non-pregnant women with low back pain will enter the study. Each group will receive two different interventions, one consisting of visual feedback when performing 10 repetitions of low back flexion, extension and right and left side-flexion and another intervention consisting of the same low back movements without visual feedback. Participants will be assessed for pain intensity, pain location, disability, kinesiophobia, catastrophizing, perception of the low back, flexion range of motion and time to perform the sit to stand test both at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The sample will consist of 15 pregnant participants (ideally between the 2nd and 3rd trimester of gestation) with chronic idiopathic low back pain and a group of 15 non-pregnant women with chronic idiopathic low back pain.

Exclusion Criteria:

* Pregnant women with risk pregnancy will be excluded as well as low back pain with a known cause (e.g. radiculopathy) and all participants with serious pathologies (e.g. history of trauma, surgery for less than 12 months, neurological pathologies, tumors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  Measured using the visual analogue scale, which measures pain intensity (range: 0-10 and higher values are indicative of higher pain intensity)
Pain intensity | Immediately after the intervention (at 30 minutes)
  Measured using the visual analogue scale, which measures pain intensity (range: 0-10 and higher values are indicative of higher pain intensity)

SECONDARY OUTCOMES:
Pain location | Baseline
  Measured using a body chart
Pain location | Immediately after the intervention (at 30 minutes)
  Measured using a body chart
Disability | Baseline
  Assessed using the Roland Morris Questionnaire, which assesses low back pain associated disability (range: 0-24 and higher values indicate higher disability)
Disability | Immediately after the intervention (at 30 minutes)
  Assessed using the Roland Morris Questionnaire, which assesses low back pain associated disability (range: 0-24 and higher values indicate higher disability)
Catastrophizing | Baseline
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Catastrophizing | Immediately after the intervention (at 30 minutes)
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Low back perception | Baseline
  Assessed by asking participants to draw how they perceive their low back to be
Low back perception | Immediately after the intervention (at 30 minutes)
  Assessed by asking participants to draw how they perceive their low back to be
Flexion range of motion | Baseline
  The distance between the 3rd finger and the floor is measured with a ruler when participants lean forward.
Flexion range of motion | Immediately after the intervention (at 30 minutes)
  The distance between the 3rd finger and the floor is measured with a ruler when participants lean forward.
Time taken to sit and stand 5 times | Baseline
  Measured using the sit-to-stand test, i.e., the time, in seconds, that a participant takes to sit and stand from a common chair 5 consecutive times.
Time taken to sit and stand 5 times | Immediately after the intervention (at 30 minutes)
  Measured using the sit-to-stand test, i.e., the time, in seconds, that a participant takes to sit and stand from a common chair 5 consecutive times.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Principal Investigator — Aveiro University
Locations (1):
- Escola Superior de Saúde, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No